CLINICAL TRIAL: NCT06294236
Title: A Phase 1 Study Evaluating SC291, a Hypoimmune, Allogeneic CD19-directed CAR T Cell Therapy, in Subjects With Severe Relapsed or Refractory Autoimmune Diseases (GLEAM)
Brief Title: Study Evaluating SC291 in Subjects With Severe r/r B-cell Mediated Autoimmune Diseases (GLEAM)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sana Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SC291-102
Record Dates: First submitted 2024-02-12; First posted 2024-03-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lupus Erythematosus; Systemic Lupus Erythematosus; SLE (Systemic Lupus); Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatous Polyangiitis; Microscopic Polyangiitis
Keywords: Autoimmune Disease; Systemic Lupus Erythematosus; Lupus Nephritis; Lupus; Extrarenal Lupus; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatous Polyangitis; Microscopic Polyangiitis; CAR T Cell Therapy; Allogeneic; Hypoimmune; CD19; Cyclophosphamide; Fludarabine; Cellular Therapy; SC291; ANCA Associated Vasculitis; SLE; ANCA; Vasculitis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Autoimmune Diseases; Lupus Nephritis; Vasculitis | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LN Cohort (Experimental): SC291 with lymphodepleting therapy
  Interventions: Biological: SC291
- ERL Cohort (Experimental): SC291 with lymphodepleting therapy
  Interventions: Biological: SC291
- AAV Cohort (Experimental): SC291 with lymphodepleting therapy
  Interventions: Biological: SC291

INTERVENTIONS:
Biological: SC291 — SC291 is an allogeneic CAR T cell therapy
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
SC291-102 is a Phase 1 study to evaluate SC291 safety and tolerability, preliminary clinical response, cellular kinetics and exploratory assessments for subjects with severe autoimmune diseases.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease with multisystemic organ involvement that is often fatal. SLE is subcategorized as extrarenal lupus (ERL) or lupus nephritis (LN). B cell depletion therapies have played an important role in the treatment of multiple B cell-driven autoimmune diseases.

Subjects included in this trial will be subjects with diagnoses of systemic lupus erythematosus (SLE) including lupus nephritis (LN) and extrarenal systemic lupus erythematosus (ERL), or anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV) (including Granulomatous Polyangitis and Microscopic Polyangiitis) who have refractory disease, have relapsed and have not shown appropriate clinical responses following prior systemic treatments.

This study is being conducted to evaluate the safety and efficacy of an investigational cell therapy, SC291, that can be given to patients with LN, ERL or AAV, in separate parallel cohorts, who have active disease.

A single dose of SC291 will be evaluated in patients who are pretreated with a standard regimen including cyclophosphamide (CY) and fludarabine (FLU).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75
2. For LN cohort:

   * Diagnosis of SLE based on the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR)
   * Biopsy-proven LN class III or IV, according to 2018 Revised International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria
   * Refractory disease to ≥ 2 prior treatment regimens
3. For ERL cohort:

   * Diagnosis of SLE based on the 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for adult SLE
   * Severe or relapsing disease not responding to at least 2 prior recent disease-modifying therapies
4. For AAV Cohort, diagnosed with Granulomatous Polyangiitis (GPA) or Microscopic Polyangiitis (MPA) based on the 2022 ACR/EULAR classification criteria

Exclusion Criteria:

1. Prior CD19-directed cell therapy including CAR T treatment or other genetically modified cell therapy (e.g., Natural Killer (NK) cell)
2. For LN and ERL Cohorts, central nervous system (CNS) lupus manifestations or history or presence of CNS disorder
3. For LN and ERL Cohorts, diagnosis of anti-phospholipid antibody syndrome
4. For AAV Cohort only, Diagnosis of Eosinophilic Granulomatosis with Polyangiitis (EGPA) as defined by the 2022 ACR/EULAR classification criteria for EGPA -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability of SC291 | 24 months
  Safety and Tolerability: Proportion of subjects experiencing adverse events and dose-limiting toxicities

SECONDARY OUTCOMES:
Evaluate preliminary clinical response to SC291 | 12 months
  Change from baseline in renal function as measured by Estimated Glomerular Filtration Rate (eGFR) (calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)
Evaluate preliminary clinical response to SC291 | 12 months
  Change from baseline in proteinuria as measured by Urine Protein Creatinine Ratio (UPCR)
Evaluate preliminary clinical response to SC291 | 12 months
  Duration of drug free remission
Evaluate preliminary clinical response to SC291 | 12 months
  Time to relapse
Evaluate preliminary clinical response to SC291 (LN and ERL Cohorts) | 12 months
  Change from baseline of Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K)
Evaluate preliminary clinical response to SC291 (LN Cohort) | 12 months
  Change in disease activity as measured by proportion of subjects achieving complete renal response or partial renal response
Evaluate preliminary clinical response to SC291 (ERL Cohort) | 12 months
  Change in disease activity as measured by proportion of subjects achieving modified Definitions Of Remission In Systemic Lupus Erythematosus (DORIS) remission
Evaluate preliminary clinical response to SC291 (AAV Cohort) | 12 months
  Change in disease activity as measured by proportion of subjects achieving remission (Birmingham Vasculitis Activity Score version 3 [BVAS v3] of 0)
Evaluate preliminary clinical response to SC291 (AAV Cohort) | 12 months
  Change in disease activity as measured by change from baseline in BVAS v3
Evaluate cellular kinetics and persistence of SC291 | 24 months
  Levels of SC291 CAR+ T cells in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Lee, Study Director — Sana Biotechnology, Inc.
Locations (5):
- United States (5):
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Swedish Medical Center, Seattle, Washington